CLINICAL TRIAL: NCT03802643
Title: Assessment of Oxygenation Values Before General Anesthesia in Elective Surgery
Brief Title: Preoxygenation Before General Anesthesia
Acronym: PREOX2018
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Parma (Other)
Responsible Party: Principal Investigator, Elena Giovanna Bignami, Professor, University of Parma
Other Study IDs: 530/2018/OSS/AOUPR
Record Dates: First submitted 2019-01-03; First posted 2019-01-14 (Actual); Last update posted 2019-01-14 (Actual); Status verified 2019-01

CONDITIONS: Anesthesia; Preoxygenation
Keywords: Oximetry; Desaturation of Blood; Postoperative pulmonary complications

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Week
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Rationale of the study: we aim to clarify the question (related to still unclear and not univocal response) about the protective or unnecessary role of preoxygenation in non-critically ill patients (otherwise with no high risk of desaturation) undergoing general anesthesia before elective surgery.

It will be also necessary differentiate the development of postoperative complications (pulmonary, cardiovascular, neurological, surgical) due to preoxygenation from the ones related with patient comorbidity, intraoperative and surgical causes, tube disconnection.

Procedure: patient's informed consent signature for adhesion at the study will be initially requested. With their acceptance, parameters will be recorded anonymously in the Case Report Form, identified by their initials and an alphanumeric code, until hospital discharge.

The parameters analyzed will be related to:

* preoperative evaluation; about anamnesis, health general conditions, blood oxygen saturation (Sat02), Metabolic Equivalent of Task (METs)
* intraoperative evaluation; about oxygenations values, recorded before/during induction and maintenance of general anesthesia
* postoperative evaluation; about postoperative complications, pulmonary primarily, and secondary cardiovascular, neurological and surgical, based on the medical record.

The data wil be transferred on Excel worksheet, utilized for descriptive analysis related at every variable. By multivariate logistic regression will be evaluated the major factors influencing postoperative pulmonary complications (PPCs) onset in patients undergoing preoxygenation for elective surgery

DETAILED DESCRIPTION:
Background of the study:

Preoxygenation is a widely used technique that improves the safety of endotracheal intubation. The procedure is carried out by supplying 100% oxygen (FiO2 of 1.0) before the induction of general anesthesia until both end-tidal oxygen (EtO2)>90% and end-tidal N2 (EtN2)<5% are reached. Both these markers define the efficacy of the procedure. As a result, the lung oxygen content is increased far beyond normal oxygen consumption by saturating the functional residual capacity with 100% oxygen. This allows for a longer safe apnea time (i.e. the time required for oxyhemoglobin saturation to drop below 90%). The rate at which oxyhemoglobin saturation drops during apnea indicates the efficiency of the maneuver.

This procedure is strongly recommended for all patients undergoing general anesthesia since it lengthens safe laryngoscopy time and grants a wider timeframe to respond to a "cannot intubate/cannot oxygenate" (CICO) scenario, a rare yet life threatening situation. It remains unclear whether this should be considered mandatory for non-critically ill and non-obese patients since their oxygen reserves should suffice for the time required to perform endotracheal intubation or regain spontaneous breathing in the event of a CICO scenario. Nonetheless, the guidelines for the management of endotracheal intubation, proposed by the Difficult Airway Society in 2015 United Kingdom state how it is pivotal to preoxygenate every patient before attempting to intubate. Several methods of preoxygenation have been validated and compared according to duration of safe apnea time, duration of the procedure, success rate (defined as "avoiding manual re-ventilation"), and patient tolerance. The choice between these techniques is based on patient characteristics (age, sex, Body Mass Index, American Society of Anesthesiologist score, Cormack-Lehane grade and Glasgow Coma Scale), settings (e.g., operating room, Intensive Care Unit, emergency situations), equipment, and anesthesiologist's preferences. The two standard approaches are six deep breaths in 1 min and tidal volume breathing for three to 5 min, both at 100% inspired oxygen via a face mask.

The main side effect of preoxygenation is absorption atelectasis that occurs when delivering 100% inspired oxygen. This can be avoided using a lower inspired oxygen concentration (90%), positive pressure techniques, and/or recruitment maneuvers post-endotracheal intubation. Due to the short duration of the procedure, the production of reactive oxygen species and cardiovascular responses are minimal and should not prevent routine preoxygenation.

ELIGIBILITY:
Inclusion Criteria:

* informed consent signature
* eligible for preoxygenation before general anesthesia, in elective surgery
* age > 18 years
* surgery duration > 30 min

Exclusion Criteria:

* emergency/urgent surgery
* severe respiratory disease: Chronic Obstructive Pulmonary Disease stages III-IV, pulmonary fibrosis, documented bullous emphysema, severe emphysema, pneumothorax
* uncontrolled asthma
* severe cardiac disease: Heart Failure stages III-IV (New York Heart Association), coronary artery disease stages III-IV (Canadian Cardiovascular Society)
* previous thoracic surgery
* pregnancy (excluded by anamnesis or laboratory test)
* informed consent refusal

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Non-critically ill patients (with no high risk of desaturation) undergoing general anesthesia before elective surgery.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2018-12-20 (Actual); Primary Completion 2019-12-20 (Estimated); Study Completion 2020-01-20 (Estimated)

PRIMARY OUTCOMES:
Evaluation of preoxygenation use in elective surgery, reporting oxygenations values | From before induction of general anesthesia until the end of surgical procedure, up to 10 hours
  Assessment of its efficacy and efficiency in non-critically ill patients, reporting blood oxygen levels just before induction, during induction and maintenance of general anesthesia
Incidence of postoperative pulmonary complications (PPC) related to preoxygenation | From immediately after surgery until hospital discharge, up to 26 weeks
  Differentiating PPCs due to preoxygenation from the ones related with patient comorbidity, intraoperative and surgical causes, tube disconnection

SECONDARY OUTCOMES:
Incidence of intraoperative desaturation/hypoxia | From achieved endotracheal intubation until the end of surgical procedure, up to 10 hours
Incidence of cardiovascular postoperative complications | From immediately after surgery until hospital discharge, up to 26 weeks
Incidence of neurological postoperative complications | From immediately after surgery until hospital discharge, up to 26 weeks
Incidence of surgical postoperative complications | From immediately after surgery until hospital discharge, up to 26 weeks
Incidence of Intensive Care Unit admission and its duration | From immediately after surgery until hospital discharge, up to 26 weeks
Incidence of length of in-hospital stay | From immediately after surgery until hospital discharge, up to 26 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Michela Tosi, MD, Principal Investigator — Azienda Ospedaliero-Universitaria di Parma; Benedetta Siroli, MD, Principal Investigator — University of Parma; Samantha Gorgoglione, MD, Principal Investigator — University of Parma; Valentina Bellini, MD, Principal Investigator — University of Parma; Leonardo Fortunati, MD, Principal Investigator — University of Parma; Andrea Parodi, MD, Principal Investigator — University of Parma; Andrea Briolini, MD, Principal Investigator — University of Parma
Locations (1):
- Azienda Ospedaliero-Universitaria di Parma, Parma, Italy